CLINICAL TRIAL: NCT04028011
Title: Evaluación clínica de Una tecnología Ambulatoria Para diagnóstico Del sueño
Brief Title: Clinical Evaluation of a Wearable Technology for the Diagnosis of Sleep Apnoea
Status: Recruiting | Type: Observational
Sponsor: Acurable Ltd. (Industry)
Collaborators: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Sponsor
Other Study IDs: 720/19/EC
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PSG and novel wearable device: 75 patients will wear polysomnography at the same time as the Novel wearable device
  Interventions: Diagnostic Test: Novel Wearable device
- PG and novel wearable device: 75 patients will wear polygraphy at the same time as the novel wearable device
  Interventions: Diagnostic Test: Novel Wearable device

INTERVENTIONS:
Diagnostic Test: Novel Wearable device — patient will wear novel wearable device overnight along with normal standard of care

SUMMARY:
This trial will aim to test a new wearable device for the diagnosis of Sleep Apnoea.

DETAILED DESCRIPTION:
This clinical trial will test a new wearable device for the diagnosis of Sleep Apnoea against Multi-channel polygraphy and Polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been referred to a sleep clinic due to suspicion of sleep apnoea.
* patients between the age of 18 yo and 80 yo

Exclusion Criteria:

* who are not fluent in Spanish, or who have special communication needs.
* Known allergy to the adhesive dressing.
* patients with physical or mental impairments who would not be able to use the new technology on their own.
* patients with very loose/saggy skin in the neck area which would unavoidably result on AcuPebble swinging if moving the neck.
* patients with pacemakers or who have any type of implanted electronic device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred for suspicion of sleep apnoea
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivities and Specificity for diagnosis of sleep apnoea studies with novel wearable device | 6 months
  The study aims to compare the diagnosis result of the novel wearable device against standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Fernando Sanchez Gomez, MD, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Virgen Macarena Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: No